CLINICAL TRIAL: NCT05067088
Title: Novel physIologiC prEdictors of Positive Airway Pressure Effectiveness: NICEPAP Study Prospective Cohort
Brief Title: Novel physIologiC prEdictors of Positive Airway Pressure Effectiveness
Acronym: NICEPAP
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000024615; 1K23HL159259-01 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Continuous positive airway pressure (CPAP); Physiologic sleep apnea traits (endotypes); CPAP adherence; CPAP efficacy; Patient-centered sleep apnea outcomes; Precision medicine; Arousal threshold; Loop gain; Pharyngeal collapsibility; Pharyngeal muscle compensation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CPAP (all patients receive CPAP as part of routine clinical care) — Continuous positive airway pressure
  Other Names: Exposure: arousal threshold; Exposure: loop gain; Exposure: pharyngeal collapsibility; Exposure: pharyngeal muscle compensation

SUMMARY:
Millions of Americans suffer from high blood pressure, diabetes, strokes and motor vehicle accidents due to ineffective treatment of obstructive sleep apnea (OSA). Our preliminary data suggest that physiological causes of OSA such as easy arousability (low arousal threshold) or unstable breathing control (high loop gain) may influence effectiveness of OSA's most common treatment, continuous positive airway pressure (CPAP). The NICE-PAP study will examine how the physiologic traits that cause OSA in each individual impact CPAP effectiveness and can lead to personalized OSA treatments that improve patient lives.

DETAILED DESCRIPTION:
Most patients with OSA who are prescribed the gold-standard therapy, CPAP, are ineffectively treated. This is due to 1) poor CPAP adherence, 2) high residual apnea in 20% of users (low efficacy) and 3) inconsistent symptom improvement. To improve CPAP effectiveness, we propose to address novel physiologic targets that cause OSA in each individual: arousability (arousal threshold), ventilatory control sensitivity (loop gain) and pharyngeal muscle compensation.

Our overall objective is to determine the contribution of these traits to CPAP effectiveness independently of established biological, psychological and social predictors. This study leverages state-of-the art sleep study analysis tools and validated measures of the determinants of CPAP effectiveness to create a pragmatic, prospective cohort (n=267) of OSA patients. This unique dataset will help determine whether physiologic causes of OSA influence CPAP adherence, efficacy, sleep quality, symptoms, function and quality of life. The results will inform design and conduct of a randomized clinical trial designed to modify physiologic traits such as easy arousability to improve CPAP effectiveness and other patient-centered outcomes in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age of >18 years
2. Newly diagnosed OSA naïve to CPAP
3. Apnea hypopnea index (AHI) ≥5/hr on in-laboratory polysomnography or home sleep test acquired and scored using standard criteria(59)
4. Referred for CPAP adherence management at Yale New Haven Hospital Sleep Center

Exclusion Criteria:

1. Need for supplemental oxygen
2. Central apnea index comprising >50% of the AHI
3. Treatment recommendation with another modality (e.g., Bilevel PAP, Adaptive Servo-Ventilation, Automatic Volume Pressure Assured Pressure Support)
4. A referral for a sleep disorder other than OSA (i.e., narcolepsy, sleep related movement disorder, circadian rhythm sleep-wake disorder)
5. Prior CPAP or Auto-CPAP use over the past 3 years
6. Unstable medical or mental health condition (e.g., decompensated heart failure, end-stage chronic obstructive pulmonary disease, end stage renal disease, psychosis)
7. Inability to participate in the informed consent process (e.g., cognitive impairment)
8. Pregnancy
9. Non-English language use as only means of communication (because the research budget does not provide adequate resources to ensure that the needs of non-English speaking patients can be adequately addressed)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be drawn from the clinical population of patients referred for evaluation to the Yale New Haven Hospital Sleep Center. Currently, 38% of patients at YNHH with diagnosis of OSA are women, 65% are White, 12% Black, 10% Hispanic, 1% Asian, 1% Pacific Islander and remainder selecting other or unknown classification. We expect a similar proportion of enrolled subjects. Inclusion of vulnerable population subjects such prisoners or institutionalized individuals will be rare as these patients are infrequently evaluated sleep medicine clinics, however, they will not be excluded. Subjects who are undocumented immigrants to the U.S. will not be excluded and will undergo an informed consent process individualized in each encounter. Inclusion/exclusion criteria are noted above.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
CPAP adherence | 6 months
  average daily CPAP use (hours/night)
CPAP efficacy | 6 months
  average daily residual apnea hypopnea index on CPAP (events/hour)
OSA related quality of life measured by Functional Outcomes of Sleep Questionnaire (FOSQ) short form | 6 months
  FOSQ short form average scores, Range 0 - 5, higher scores reflect worse quality of life and function.

SECONDARY OUTCOMES:
CPAP adherence (dichotomous) | 3 months
  dichotomized measure of >4 hours/night for >70% of nights
CPAP adherence | 1 month
  average daily CPAP use (hours/night)
CPAP adherence | 12 months
  average daily CPAP use (hours/night)
CPAP efficacy (dichotomous) | 6 months
  residual AHI >=10/hour
Sleep quality: Patient-Reported Outcomes Measurement Information System (PROMIS) scores | 6 months
  PROMIS scores, Range 0 - 40, higher scores reflect worse quality
Sleep related impairment: Patient-Reported Outcomes Measurement Information System (PROMIS) scores | 6 months
  PROMIS - impairment scores, range 0 - 40, higher scores reflect greater impairment
Insomnia: Insomnia Severity Index (ISI) | 6 months
  ISI scores, Range 0 - 28; higher scores reflect higher insomnia burden/severity
Epworth sleepiness scale | 6 months
  Epworth sleepiness scale scores, Range 0 - 24; higher scores signify greater sleepiness
Anxiety: Hospital Anxiety and Depression Scale - Anxiety subscale scores | 6 months
  Hospital Anxiety and Depression Scale - Anxiety subscale scores range 0 - 21; higher scores signify greater anxiety symptoms
Depression: Hospital Anxiety and Depression Scale - Depression subscale scores | 6 months
  Hospital Anxiety and Depression Scale - Depression subscale scores, Range 0 - 21; higher scores signify greater depression symptoms
Attention | 6 months
  median reaction time and mean slowest 10% reaction time from a 5-min smartphone-based psychomotor vigilance test.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Zinchuk, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Sleep Center, North Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zinchuk A, Edwards BA, Jeon S, Koo BB, Concato J, Sands S, Wellman A, Yaggi HK. Prevalence, Associated Clinical Features, and Impact on Continuous Positive Airway Pressure Use of a Low Respiratory Arousal Threshold Among Male United States Veterans With Obstructive Sleep Apnea. J Clin Sleep Med. 2018 May 15;14(5):809-817. doi: 10.5664/jcsm.7112. PMID 29734986
- [Background] Zinchuk AV, Redeker NS, Chu JH, Liang J, Stepnowsky C, Brandt CA, Bravata DM, Wellman A, Sands SA, Yaggi HK. Physiological Traits and Adherence to Obstructive Sleep Apnea Treatment in Patients with Stroke. Am J Respir Crit Care Med. 2020 Jun 15;201(12):1568-1572. doi: 10.1164/rccm.201911-2203LE. No abstract available. PMID 32083949
- [Background] Zinchuk AV, Chu JH, Liang J, Celik Y, Op de Beeck S, Redeker NS, Wellman A, Yaggi HK, Peker Y, Sands SA. Physiological Traits and Adherence to Sleep Apnea Therapy in Individuals with Coronary Artery Disease. Am J Respir Crit Care Med. 2021 Sep 15;204(6):703-712. doi: 10.1164/rccm.202101-0055OC. PMID 34156917
- [Derived] Anwar AI, Byrne S, Sharma A, Sands S, Wellman A, Redeker NS, Yaggi H, Zinchuk AV. Novel physiologic predictors of positive airway pressure effectiveness (NICEPAP) study: rationale, design and methods. Sleep Breath. 2024 Oct;28(5):2005-2015. doi: 10.1007/s11325-024-03099-w. Epub 2024 Jul 12. PMID 38995327